CLINICAL TRIAL: NCT07297277
Title: An Observational Cross-Sectional Blind Comparison to Evaluate the Level of Agreement Between AAMI/ESH/ISO Universal Standard Requirements and the HUAWEI D2 Watch-Type Wrist Blood Pressure Monitor
Brief Title: Evaluating the Level of Agreement Between AAMI/ESH/ISO Universal Standard Requirements and the HUAWEI D2 Watch-Type Wrist Blood Pressure Monitor
Status: Recruiting | Type: Observational
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Other Study IDs: 10374
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-10

CONDITIONS: Blood Pressure Monitoring
Keywords: Blood Pressure; Auscultatory; Oscillometric; Watch Type Monitor; Validation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Pressure Measurements: All participants will have blood pressure measurements taken in accordance with the AAMI/ESH/ISO validation guidelines.
  Blood pressure cuff placed on upper arm and HAUWEI D2 watch placed on wrist of same arm.
  Participants seated in silence for at least 5 minutes. Two observers will undertake reference BP measurements simultaneously, blinded to each other's measurements.
  Same arm sequential method of testing with a 60-second rest between each measurement as follows:
  Baseline BP: reference BP measurement/test device BP measurement.
  Validation BP measurements for accuracy evaluation: 1st reference BP measurement;1st test device measurement; 2nd reference BP measurement; 2nd test device measurement; 3rd reference BP measurement; 3rd test device measurement; 4th reference BP measurement.
  If there is observer disagreement >4mmHg in Systolic or Diastolic for reference BP then another pair of BP readings (test and reference) is taken up to a maximum of 8 pairs.

SUMMARY:
Getting an accurate blood pressure (BP) reading is essential for diagnosing high blood pressure and managing it effectively. High blood pressure is a major health problem, causing about 9.4 million deaths worldwide each year. More people need to monitor their BP at home, so there is greater demand for easy-to-use devices. Traditional BP monitors with arm cuffs can be bulky, uncomfortable, and awkward to use.

Modern technology has made it possible to measure BP using wearable devices like smartwatches. HUAWEI has developed a wrist watch that can measure BP and has been tested to meet international standards. The watch passed these tests and was approved for people to use at home to check their own BP. However, the HUAWEI watch was only tested on people in China and the investigators need to know if it works for people from other countries and ethnic backgrounds.

DETAILED DESCRIPTION:
Accurate measurement of blood pressure (BP) is a necessity for the reliable diagnosis and proficient management of hypertension. However, validation of blood pressure monitoring devices only began in the 1980's, followed by a series of ad-hoc validation protocols from differing organisations such as the Advancement of Medical Instrumentation (AAMI), the British Hypertension Society (BHS), the German Hypertension League, the European Society of Hypertension (ESH), and the International Organisation for Standardization (ISO) over the subsequent three decades. The need for a universally acceptable protocol was recognised and members of the AAMI, ESH, and ISO committees collaborated to re-examine the aspects of validation to achieve a consensus on an optimal validation standard.

With an increased prevalence of hypertension, causing approximately 9.4 million deaths per year worldwide, the demand for non-invasive arterial pressure monitoring devices has also increased to help patients manage blood pressure (BP). Traditionally, non-invasive BP measurement techniques include auscultatory and oscillometric devices, however, these can present with several limitations in terms of cuff size, instruments' bulky volume, and discomfort caused by external pressure. Advancements in technology has meant that wearable devices are becoming readily available for various health related measurements, including BP. The HUAWEI Technology have developed an automated oscillometric wearable wrist watch-type device for BP measurement that has recently been validated in accordance with the AAMI/ESH/ISO Universal Standard requirements and can be recommended for self-measurement. However, while this research concluded the HUAWEI watch fulfilled the requirements for self-measurement in the general population, it should be noted that the study was conducted within the Chinese population only. Consequently, to ensure generalisation to a wider population, it is important to examine the HUAWEI watch validity within differing populations. Therefore, the aim of this study will be to explore if the HUAWEI D2 watch-type blood pressure monitor meets the AAMI/ESH/ISO Universal Standard requirements in differing populations.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Written informed consent provided

Exclusion Criteria:

* Cardiac Arrythmias
* Peripheral Arterial Disease
* Known Heart Disease
* Pregnancy
* Diagnosis of Secondary Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample with normotensive, pre-hypertensive, and hypertensive blood pressure values recruited from diverse ethnic populations in the Tyne and Wear area.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Level of Agreement Between Auscultatory and HUAWEI D2 Watch Blood Pressure Measurements. | Baseline
  The level of agreement between auscultatory systolic blood pressure (mmHg) and diastolic blood pressure (mmHg), and the HUAWEI D2 watch systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) measurements will be determined using the AAMI/ESH/ISO standard requirements for blood pressure device validation.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Cucato, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min S, Kim DH, Joe DJ, Kim BW, Jung YH, Lee JH, Lee BY, Doh I, An J, Youn YN, Joung B, Yoo CD, Ahn HS, Lee KJ. Clinical Validation of a Wearable Piezoelectric Blood-Pressure Sensor for Continuous Health Monitoring. Adv Mater. 2023 Jun;35(26):e2301627. doi: 10.1002/adma.202301627. Epub 2023 May 11. PMID 36960816
- [Background] Zhang W, Zhou YN, Zhou Y, Wang JG. Validation of the watch-type HUAWEI WATCH D oscillometric wrist blood pressure monitor in adult Chinese. Blood Press Monit. 2022 Oct 1;27(5):353-356. doi: 10.1097/MBP.0000000000000608. Epub 2022 May 27. PMID 35687029
- [Background] O'Brien E, Atkins N. State-of-the-market from the dableducational.org website. Blood Press Monit. 2007 Dec;12(6):377-9. doi: 10.1097/MBP.0b013e328244de94. PMID 18277314
- [Background] Stergiou GS, Palatini P, Asmar R, Ioannidis JP, Kollias A, Lacy P, McManus RJ, Myers MG, Parati G, Shennan A, Wang J, O'Brien E; European Society of Hypertension Working Group on Blood Pressure Monitoring. Recommendations and Practical Guidance for performing and reporting validation studies according to the Universal Standard for the validation of blood pressure measuring devices by the Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO). J Hypertens. 2019 Mar;37(3):459-466. doi: 10.1097/HJH.0000000000002039. PMID 30702492